CLINICAL TRIAL: NCT03017859
Title: High Flow Nasal Cannula as a Treatment for Obstructive Sleep Apnea
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rabin Medical Center (Other)
Responsible Party: Principal Investigator, Mordechai Kremer, Head of Pulmonary Institute, Rabin Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RMC-16-0152
Record Dates: First submitted 2017-01-09; First posted 2017-01-11 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2017-01

CONDITIONS: Sleep Apnea, Obstructive
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- High flow nasal cannula treatment (Experimental): Airvo 2 device will be used to administer high flow air during the night
  Interventions: Device: High flow nasal cannula

INTERVENTIONS:
Device: High flow nasal cannula — We shall use the Airvo 2 device to administer humidified and warmed air at high flow during sleep.

SUMMARY:
A single center, prospective study to assess the efficacy of high flow nasal cannula (HFNC) in improving obstructive sleep apnea (OSA) parameters in patients with reduced tolerance to continuous positive airway pressure (CPAP) treatment.

DETAILED DESCRIPTION:
A single center, prospective study. The study would include 30 patients diagnosed within the past 2 years with moderate to severe OSA (AHI>=15) at the Rabin Medical Center (RMC) sleep lab, and who are intolerant to CPAP treatment. Following signing an informed consent form, these patients would undergo polysomnography (PSG) while treated with HFNC. The HFNC PSG outcome measures will be compared to the baseline PSG done within the past 2 years and to an additional PSG while connected to a CPAP device.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years
* Confirmed diagnosis of obstructive sleep apnea, diagnosed at RMC sleep lab in the past 2 years
* Apnea Hypopnea Index (AHI)≥15
* Patient has difficulties to adjust or comply with CPAP treatment
* Signed Informed Consent Form

Exclusion Criteria:

* Patients who need bilevel positive airway pressure (BIPAP)
* Known carbon dioxide (CO2) retainers
* Weight change>10% compared to time of OSA diagnosis
* Clinically unstable patients
* Pregnant women or special populations (e.g. children or patients unable to give informed consent)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-01; Primary Completion 2018-07 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Apnea Hypopnea Index (AHI) | During at least 2 hours of sleep time
  Comparison of HFNC AHI to baseline AHI and to CPAP AHI

SECONDARY OUTCOMES:
Percent of hypoxemia time | During at least 2 hours of sleep time
  O2 saturation (SO2)<90% as measured by pulse oximeter
Minimal SO2% | During at least 2 hours of sleep time
Adverse events reported while using HFNC | During at least 2 hours of sleep time
Sleep efficiency | During at least 2 hours of sleep time
Total sleep time | During at least 2 hours of sleep time

OTHER OUTCOMES:
Percent rapid eye movement (REM) sleep | During at least 2 hours of sleep time
Percent Deep sleep | During at least 2 hours of sleep time
User experience with HFNC | During at least 2 hours of sleep time
  To be assessed in the following morning with questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Mordechai R Kramer, MD, Principal Investigator — Pulmonary Institute, Rabin Medical Center, Israel

IPD SHARING:
Plan to Share IPD: No